CLINICAL TRIAL: NCT06933095
Title: Optimizing CNS DHA Delivery in Elderly Adults at Risk for Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert McNamara, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CNS DHA Delivery
Record Dates: First submitted 2024-12-04; First posted 2025-04-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Eldery People; Cognitive Decline; Memory Decline; DHA CNS Delivery
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (mixture of olive oil, corn oil, palm oil) (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: LPC-EPA+DHA capsules containing omega-3 fatty acids EPA and DHA esterified to lysophosphatidylcholine (LPC-EPA+DHA)(Trade name: Lysoveta)
- fish oil (Active Comparator): Fish Oil
  Interventions: Dietary Supplement: LPC-EPA+DHA capsules containing omega-3 fatty acids EPA and DHA esterified to lysophosphatidylcholine (LPC-EPA+DHA)(Trade name: Lysoveta)
- LPC-EPA+DHA (investigational agent) capsules containing omega-3 fatty acids EPA and DHA esterified t (Experimental): LPC-EPA+DHA (investigational agent) capsules containing omega-3 fatty acids EPA and DHA esterified to lysophosphatidylcholine (LPC-EPA+DHA)(Trade name: Lysoveta)
  Interventions: Dietary Supplement: LPC-EPA+DHA capsules containing omega-3 fatty acids EPA and DHA esterified to lysophosphatidylcholine (LPC-EPA+DHA)(Trade name: Lysoveta)

INTERVENTIONS:
Dietary Supplement: LPC-EPA+DHA capsules containing omega-3 fatty acids EPA and DHA esterified to lysophosphatidylcholine (LPC-EPA+DHA)(Trade name: Lysoveta) — apsules containing omega-3 fatty acids EPA and DHA esterified to lysophosphatidylcholine (LPC-EPA+DHA)(Trade name: Lysoveta)

SUMMARY:
The purpose of this placebo-controlled trial is to compare the effects of 24-weeks supplementation with LPC-DHA and TAG-DHA on cerebrospinal fluid and blood DHA levels, as well as biomarkers of central neurodegenerative and neurotrophic activity, in elderly adults experiencing early signs of cognitive/memory decline including those with mild cognitive impairment (MCI). Extant evidence supports our overarching hypothesis that LPC-DHA supplementation will be more effective than TAG-DHA for increasing central (CSF) DHA levels and improving biomarker profiles in elderly adults. To assess this hypothesis, the following aims are proposed:

SPECIFIC AIM 1: To compare the effects of LPC-DHA and TAG-DHA supplementation on peripheral and CSF DHA levels in elderly adults experiencing early signs of cognitive/memory decline.

SPECIFIC AIM 2: To compare the effects of LPC-DHA and TAG-DHA supplementation on neurotrophic and neurodegenerative biomarkers.

Secondary Aim: To investigate whether changes in CSF DHA levels correlate with changes in objective measures of executive functioning and episodic memory performance.

ELIGIBILITY:
Inclusion Criteria:

1. men and women 55 to 82 years old;
2. presence of subjective cognitive decline or mild cognitive decline using the SCD questionnaire, DEX, EMQ, MoCA; and mCDR;
3. No contraindication to a lumbar puncture (LP) unless opting to not have the LP (e.g., thrombocytopenia, coagulopathy, concomitant use of anticoagulant medications, etc.);
4. fluency in English;
5. ability to comprehend and comply with the research protocol; and
6. provision of written informed consent.

Exclusion Criteria:

1. diagnosis of dementia due to AD, Parkinson's disease, frontotemporal dementia, multi-infarct dementia, head trauma with loss of consciousness lasting more than 5 minutes and resulting in persisting functional decline within the three years prior to enrollment, epilepsy, leukoencephalopathy, other neurological conditions that would interfere the study objectives, mMIST <8 or MoCA-MI score <7;
2. self-reported history of any psychotic disorder or bipolar disorder;
3. diagnosis of atrial fibrillation, pancreatic, liver, kidney or hematological coagulation disorder;
4. allergy to shellfish or seafood;
5. current substance use causing physiological dependence or persisting change in functional capability;
6. concomitant, regular use of medications that might affect primary outcome measures or adversely interact with the study product including anticoagulant medications;
7. weekly fish consumption more than 1 x 3 oz servings and/or use of DHA-containing supplements within 3 months prior to screening.

Ages: 55 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2029-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
CSF Docosahexaenoic acid (DHA) levels | From baseline through week 24
  Baseline-Endpoint change in CSF docosahexaenoic acid (DHA) composition (g/100 g).

SECONDARY OUTCOMES:
Amyloid-β1-42 (Aβ42) | Baseline through week 24
  Baseline-Endpoint change in blood and CSF amyloid-β1-42 concentrations (ng/ml)
Phospho-tau217 (p-tau217) | Baseline and Week 24
  Baseline-Endpoint change in blood and CSF p-tau217 concentrations (ng/ml)
Brain-derived neurotrophic factor (BDNF) | Baseline and Week 24
  Baseline-Endpoint change in blood and CSF BDNF concentrations (ng/ml)
Genotyping | Baseline
  APOE alleles (ε2, ε3, ε4) allele frequency
California Verbal Learning Test | Baseline, Week 12, Week 24
  Objective assessment of episodic memory performance (Units on a scale) Scores range from 0 to 16 for individual learning trials, 0 to 80 for total words recalled across all trials, 0 to 16 for both short and long-delay free recall, and 0 to 16 for total hits. Higher scores indicate better performance on verbal memory
Trail-Making Test, part B | Baseline, week 12, and week 24
  Objective measure of speed of processing/executive functioning (Units on a scale). Scores range from 0 to 300 seconds to complete the task. Lower scores indicate better performance on executive function.
Geriatric Depression Scale | Screening, Baseline, week 12, and week 24
  Assessment of depression symptom severity (Units on a scale). The score range is from 0 to 15, with higher scores indicating more severe depression.

OTHER OUTCOMES:
Blood glucose levels | Baseline, week 12, and week 24
  Fasting blood glucose concentrations (mg/dL) as a measure of glucose regulation and insulin resistance.
Blood insulin levels | Baseline, Week 12, week 24
  Fasting blood insulin concentrations (pmol/L) as a measure of glucose homeostasis and insulin effectiveness.
Blood triglycerides levels | Baseline, week 12, and week 24
  Fasting blood triglycerides concentrations (mg/dL)
Blood cholesterol levels | Baseline, week 12, and week 24
  Fasting blood cholesterol concentrations (mg/dL)
Blood alanine transaminase (ALT) levels | Baseline, week 12, and week 24
  Fasting blood alanine transaminase concentrations (U/L) as a measure of liver function
Blood aspartate aminotransferase (AST) levels | Baseline, week 12, and week 24
  Fasting blood aspartate aminotransferase concentrations (U/L) as a measure of liver function
Blood C-reactive protein (CRP) levels | Baseline, week 12, and week 24
  Fasting blood C-reactive protein levels concentrations (mg/dL) as a measure of systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Robert McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided